CLINICAL TRIAL: NCT06992999
Title: Psilocybin for Treatment of Obsessive Compulsive Disorder
Brief Title: Psilocybin for Treatment of OCD-2
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Francisco A Moreno (Other)
Collaborators: University of Arizona (Other)
Responsible Party: Sponsor-Investigator, Francisco A Moreno, Professor of Psychiatry, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00006264
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Obsessive - Compulsive Disorder
Keywords: obsessive compulsive disorder; OCD; psilocybin; psychedelic; psychedelic experiences
MeSH Terms: conditions — Compulsive Personality Disorder; Obsessive-Compulsive Disorder | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: Randomized, controlled trial of four sessions of psilocybin assigned to one of two dosing groups 1) low dose (10mg) 2) high dose (30mg) in a double masked fashion.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low Dose psilocybin (10mg) (Active Comparator): Subjects will receive a low dose (10mg) of psilocybin at four study drug ingesting sessions. Each drug ingestion session will be separated by three weeks.
  Interventions: Drug: Low Dose Psilocybin
- High dose psilocybin (30mg) (Active Comparator): Subjects will receive a high dose (30mg) of psilocybin at four study drug ingesting sessions. Each drug ingestion session will be separated by three weeks.
  Interventions: Drug: High Dose Psilocybin

INTERVENTIONS:
Drug: Low Dose Psilocybin — 10mg dose of psilocybin
  Arms: Low Dose psilocybin (10mg)
Drug: High Dose Psilocybin — 30mg dose of psilocybin
  Arms: High dose psilocybin (30mg)

SUMMARY:
Previous research indicates that psilocybin, a drug that changes activity in brain areas believed to be involved in obsessive-compulsive disorder (OCD), might improve treatment for, and improve lives of, people diagnosed with OCD. The investigators propose to study 20 patients with symptomatic OCD who are not taking mind altering medications or street drugs, to participate in a 12 week study. Participants will be assigned (by luck of the draw) to take low or high dose psilocybin in four dosing sessions separated by 3 weeks. Measurements for the severity of OCD, ability to function, perception of quality of life, safety and tolerability will be measured at baseline prior to drug administration, during the dosing periods, and at the end of study. Other measurements will include brain imaging via fMRI and brain tracing via electroencephalogram (EEG). The investigators believe that during medically supervised dosing sessions, both doses of psilocybin will be safe and well tolerated, and will reduce OCD symptoms. Because psilocybin is a potent drug and especially at the higher dose may induce altered states of consciousness, a thoughtfully implemented procedure for participant safety is in place. Information will be obtained to explore the effects of altered states of consciousness in the outcome of treatment and to find the mechanism of benefit.

DETAILED DESCRIPTION:
Obsessive-Compulsive Disorder (OCD) affects millions of Americans at some point during their lifetime, representing a great deal of individual suffering, social, and fiscal cost. Despite this, currently available medications fail to help as many as 40% of OCD patients, and those who respond to treatment often experience troublesome residual symptoms 4. Psilocybin holds promise as a novel approach in the treatment of OCD, supported by preliminary evidence that it achieves response and remission rates exceeding conventional interventions .

The broad long-term objectives of this research are to improve our available treatment options for OCD and advance the specific knowledge of neural mechanism explaining treatment response. Building on the investigative team's decades long work with synthetic psilocybin, data obtained during this proposed early phase clinical study may help improve the life of people affected with OCD and minimize society's burden.

The investigators propose a randomized, controlled trial of four sessions of psilocybin assigned to either low dose (10mg) or high dose (30 mg) in double masked fashion to 20 (10 per group) symptomatic and medication-free OCD patients. The study will evaluate the tolerability, safety, subjective experience, and efficacy of psilocybin for improving OCD, obtain the preliminary data needed as a pre-requisite to a larger-scale (efficacy or effectiveness) intervention study with dosing informed by this trial, and explore mechanism of anti-obsessional action.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old, and older
* Have OCD (DSM-5) based on diagnostic interview using the Structured Clinical Interview for DSM-5 Research Version (SCID).
* At least moderate severity: Yale-Brown Obsessive-Compulsive Scale (YBOCS) score ≥16.
* Failed at least one adequate trial of guideline concordant treatment.
* Considered safe for independent living
* Subjects must discontinue use of any of the following prescription or over the counter (OTC) products or nutritional supplements at least two weeks prior to initiating double-blind treatment:
* Monoamine oxidase (MAOI), UGT1A10, and UGT1A9 inhibitors
* Other active OCD treatments (cognitive behavioral therapy [CBT] or other psychotherapy; electrical or magnetic device treatments; pharmacological treatments such as antidepressant medications (e.g., SSRIs, SNRIs, MAOIs, TCAs, 5HT2 blockers, NERIs, etc.), lithium, antipsychotic drugs, 5-HT2 antagonists such as pimavanserin, and glutamatergic acting medications)

  * Note that fluoxetine must be discontinued at least 6 weeks prior to initiating double-blind treatment.
* 5HT2 agonists (e.g., efavirenz, lorcaserin), which may alter the response to psilocybin
* Serotonin-acting dietary supplements (e.g., 5-hydroxy-tryptophan, St. John's wort) due to potential for interaction with psilocybin and increased safety risks

Exclusion Criteria:

* Concurrent active substance use disorder, or a personal history of psychosis.
* History of psychosis among first degree relatives as determined by the Family Interview for Genetic Studies (FIGS) 32
* Medical illness based on physical examination and routine blood testing that may complicate cardiovascular safety or drug metabolism or excretion, such as uncontrolled hypertension, severe cardiac disease, or kidney or liver failure.
* Unstable Chronic Obstructive Pulmonary Disease (COPD) or severe sleep apnea
* Clinically significant renal or hepatic impairment, per clinical judgment of a study physician
* EKG QTc ≥ 450 msec
* Psychiatric comorbidity that may represent an acute risk to their own or other's safety.
* Subjects cannot require any sedative, narcotic, or neuroleptic medications on a regular basis. Any of these medications they have taken should have been stopped long enough in the past to allow for their elimination and safe withdrawal prior to starting administration of the study drug. The specific time required will be dependent on the medication the patient was previously receiving.
* Women who are pregnant, breastfeeding, or unwilling/unable to practice medically acceptable highly effective birth control (double barrier, oral and injectable pharmacological contraceptives) during the study.
* Suicidal behavior within the 12 months prior to enrollment, or significant risk of suicide as determined by the CSSRS items 4 (suicidal ideation with intent) and 5 (suicidal ideation with intent and plan) during screening or baseline assessment.
* Any condition for which MRI is contraindicated, at the discretion of a study investigator or the MRI technician, including: Pacemakers and defibrillators; artificial heart valves which are not MRI safe; any metal in head, spinal cord, eyes or chest; any electrical devices such as cochlear implants, nerve stimulators, deep brain stimulators, gastric pacemaker, or insulin or pain pumps; aneurysm clips; ferrous (i.e. non titanium alloy) implants in any part of the body.
* Use within the week prior to screening of drugs of abuse as listed in the current US DOJ DEA Drugs of Abuse Resource Guide, including:
* Cannabinoids (marijuana, synthetic cannabinoids)
* Simulants (amphetamine, cocaine, methamphetamine, methylphenidate, modafinil)
* Opioids (natural and synthetic),
* Sedatives (benzodiazepines, barbiturates, GHB, zolpidem, zaleplon, zopiclone)
* Hallucinogens (DMT, ibogaine, LSD, MDMA, psilocybin, psilocin, PSP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of orally administered psilocybin | 12 months
  Determine the acute safety and tolerability of orally administered psilocybin at low dose (10mg) and high dose (30mg) as measured with the Systematic Assessment for Treatment Emergent Events (SAFTEE) scale.

SECONDARY OUTCOMES:
Efficacy of oral administered psilocybin in patient with OCD | 12 months
  Determine the efficacy of two different doses (10mg and 30mg) of psilocybin as a treatment for OCD, and explore whether there may be a dose-response relationship. This will be based on the Yale-Brown Obsessive Compulsive Scale (Y-BOCS) score.

OTHER OUTCOMES:
Impact of psilocybin administration in brain function | 12 months
  Determine the impact of psilocybin administration in potential brain function OCD biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Moreno, MD, Principal Investigator — University of Arizona, College of Medicine, Tucson
Locations (1):
- University of Arizona-Tucson, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided